CLINICAL TRIAL: NCT06171477
Title: Regional Distribution of Ventilation in Different Respiratory Rates: A Study of Mechanically Ventilated Patients Undergoing Robot-assisted Laparoscopic Prostatectomy
Brief Title: Regional Distribution of Ventilation at Different Respiratory Rates
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Region Örebro County (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 281122
Record Dates: First submitted 2023-12-06; First posted 2023-12-14 (Actual); Last update posted 2024-05-03 (Actual); Status verified 2024-05

CONDITIONS: Mechanical Ventilation; Atelectasis; Distribution of Ventilation
MeSH Terms: conditions — Pulmonary Atelectasis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- 20-40-60 (Experimental)
  Interventions: Device: Ventilation 20-40-60
- 60-40-20 (Experimental)
  Interventions: Device: Ventilation 60-40-20
- 40-60-20 (Experimental)
  Interventions: Device: Ventilation 40-60-20

INTERVENTIONS:
Device: Ventilation 20-40-60 — The respiratory rate during mechanical ventilation will be altered from 20 to 40 and finally to 60 breaths per minute.
  Arms: 20-40-60
Device: Ventilation 60-40-20 — The respiratory rate during mechanical ventilation will be altered from 60 to 40 and finally to 20 breaths per minute.
  Arms: 60-40-20
Device: Ventilation 40-60-20 — The respiratory rate during mechanical ventilation will be altered from 40 to 60 and finally to 20 breaths per minute.
  Arms: 40-60-20

SUMMARY:
This study will investigate the distribution of gas during mechanical ventilation in patients undergoing robot assisted laparoscopic prostatectomy. The gas distribution of ventilation are monitored and data extracted using electric impedance tomography in different respiratory rates.

DETAILED DESCRIPTION:
Mechanical ventilation during anaesthesia and intensive care often results in an uneven gas distribution of ventilation. Patients anaesthetized for laparoscopic surgery and patients positioned i a Trendelenburg position is particularly at risk.

A less harmful mode of ventilation could possible lead to a more optimal ventilation with avoidance of ventilator induced lung injuries. The project will investigate if volume controlled ventilation with a higher respiratory frequency can be used in this purpose.

The researchers intend to investigate patients, without previously known lung disease, undergoing robot-assisted laparoscopic prostatectomy. After the patients have given informed consent, they will be included in the project. The distribution of ventilation will be monitored with electric impedance tomography (EIT). Once the patients have been anaesthetized, positioned with the head down and the surgical procedure have been started with insufflation of carbon dioxide we will start our test.

The investigators will perform three episodes of standardized ventilation with the respiratory rate (RR) of 20, 40 and 60. With a higher RR the tidal volume will be reduced tom maintain a constant inhaled minute volume. Data will be collected from the EIT-equipment, the anaesthesia machine and the monitoring system.

ELIGIBILITY:
Inclusion Criteria:

* Patients planned for robot-assisted laparoscopic prostatectomy
* > 18 years
* Consent to take part in the study

Exclusion Criteria:

* Impaired cognitive function
* Previously known lung disease
* Insufficient skills in Swedish language to understand information about the study

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 15 (Estimated)
Dates: Start 2024-05-02 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Distribution of ventilation | During the prostatectomy procedure
  Gas distribution of ventilation between different regions of interest monitored with electrical impedance tomography.

SECONDARY OUTCOMES:
Distribution of ventilation | During the prostatectomy procedure
  Gas distribution of ventilation measured as center of ventilation monitored with electrical impedance tomography.

CONTACTS AND LOCATIONS:
Overall Officials: Pether Jildenstål, PhD, Study Director — Örebro University, Sweden
Locations (1):
- Region Örebro län, Örebro, Sweden

IPD SHARING:
Plan to Share IPD: No